CLINICAL TRIAL: NCT02425267
Title: Effectiveness of a Home Telerehabilitation Program for People With Proximal Humerus Fracture Treated Conservatively: a Randomized Clinical Trial.
Brief Title: Effectiveness of a Home Telerehabilitation Program for People With Proximal Humerus Fracture
Acronym: TeleFracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Michel Tousignant, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-725
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Humeral Fractures, Proximal
Keywords: Telerehabilitation
MeSH Terms: conditions — Shoulder Fractures | interventions — Rehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telerehabilitation (Experimental): Telerehabilitation at home from a clinic
  Interventions: Other: Rehabilitation (Physiotherapy)
- Face-to-face intervention in a clinic (Active Comparator): Conventional physiotherapy
  Interventions: Other: Rehabilitation (Physiotherapy)

INTERVENTIONS:
Other: Rehabilitation (Physiotherapy) — The training program will be carried out twice a day, and at every day during the eight-week program, either by telerehabilitation or in the clinic or by autonomous unsupervised way. During weeks 1, 3 and 5, the patient will perform his/her exercises twice a week by telerehabilitation/clinic and the other without supervision. During the other weeks (2, 4, 6, 7, 8), the patient will benefit from one exercise session by telerehabilitation/clinic per week and will perform all other without supervision. Supervised sessions allow the therapist and the patient to adjust the program in case of problems and to ensure a smooth implementation of the program.

SUMMARY:
The main objective of the study is to compare the clinical effects of the innovative telerehabilitation approach (TELE group) compared to face-to-face visits to a clinic (CLINIC group) for patients treated for a proximal humerus fracture.

DETAILED DESCRIPTION:
Every year, one out of three elderly people make at least one fall, and 10% of them cause a fracture. Of these fractures, those of the proximal humerus, the forearm and the wrist count for approximately one third of total osteoporotic fractures in elderly people. Proximal humerus fractures can be treated surgically (eg: pinning, plate and screws, etc..) or conventionally by wearing a splint or a cast. Whether either of these approaches, the individual requires rehabilitation to prevent function limitations.

Among the possible reasons for the low use of rehabilitation services, there are 1) poor availability of rehabilitation services for fractures of the humerus; or 2) the difficulty of the elderly to travel to receive these services because of their precarious status. Telerehabilitation is a promising alternative approach that can help improve access to rehabilitation services once patients are discharged from hospital.

Some studies demonstrate that physiotherapy is a significant factor in the process of healing and functional recovery of a proximal humerus fracture, and that, for conservative or surgical treatment. This is showed by the good recovery of patients and by their satisfaction with the physiotherapy. In addition, since the majority of patients with a proximal humerus fracture are elderly, it becomes relevant to find a new way to offer quick service physiotherapy and simple and suitable to their condition.

The main objective of the study is to compare the clinical effects of the innovative telerehabilitation approach (TELE group) compared to face-to-face visits to a clinic (CLINIC group) for patients treated for a proximal humerus fracture.

The research hypothesis are:

1. TELE intervention will be as effective as CLINIC intervention to improve upper extremity function.
2. TELE intervention will be as effective as CLINIC intervention to improve deficiencies of the shoulder (increase range of motion).
3. Participants who received the TELE intervention will be as satisfied of their care as participants who received the CLINICL intervention.
4. TELE intervention will be less costly compared to the CLINIC intervention.

Methodology: The study has a randomized control trial design. The study population of interest is individuals who have had proximal humerus fracture and who receive a conservative treatment at the Centre Hospitalier Universitaire de Sherbrooke (CHUS) and who are returning at home. Participants will be recruited during their visit at the emergency or outpatient clinic by the medical team or research nurse assistant. The investigators expect to recruit 52 participants, that is to say 26 per group. All evaluations will be completed in the research center/hospital and will be approximately 1.5 hour in duration. The first evaluation will be conducted when medical team will ask for rehabilitation (T1) to allow participant base measures to be collected. The other evaluation will be conducted immediately after the 2-month intervention (T2). The independent variable is conventional physiotherapy and experimental intervention by telerehabilitation. The dependant variables are 1) upper extremity function; 2) range of motion; 3) user satisfaction; 4) cost of services according to the healthcare system.

Platform used: In this study, a platform based on a technological infrastructure that was developed and tested in previous telerehabilitation studies will be used. The infrastructure combines a clinical information system with videoconference components (Tandberg 550 MXP, H 264) and uses cameras that are controlled by the clinician using computer software.

The difference between the two groups will then be compared using a t-test or a chi-square test. The economic analysis will be a type of cost-effectiveness. The cost per unit of change in the main dependent variable (Constant Score) will be determined for the two groups (TELE and CONTROL) and the cost differential will be established.

ELIGIBILITY:
Inclusion Criteria:

* Proximal humerus fracture (without surgery)
* Return home after discharge from hospital
* Be able to exercise;
* Have sufficient verbal and written understanding to participate to telerehabilitation sessions, and to be able complete the questionnaires;
* Have access to high-speed Internet at home.

Exclusion Criteria:

* Presence of intra-articular type proximal humerus fracture, which can lead to a greater risk of complication and may require a longer recovery time
* Fracture surgery as a treatment
* Presence of any other type of upper body fracture which can interfere with rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01-26 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Shoulder function (score /100) | Pre-intervention: 1 to 3 weeks post fracture (T1) and Post-intervention: after the 8-week intervention (T2)
  Constant score

SECONDARY OUTCOMES:
Range of motion (degrees, measured with a goniometer) | Pre-intervention: 1 to 3 weeks post fracture (T1) and Post-intervention: after the 8-week intervention (T2)
  flexion, extension, abduction,internal and external rotation
Satisfaction with the care received (score /56) | Post-intervention: after the 8-week intervention (T2)
  Health care satisfaction questionnaire
Cost of services from the perspective of the health system | Post-intervention: after the 8-week intervention (T2)
  "Cost-analysis of telemedicine" from Minnesota University

CONTACTS AND LOCATIONS:
Overall Officials: Michel Tousignant, PT, PhD, Principal Investigator — Research Centre on Aging
Locations (1):
- Research Center on Aging, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Derived] Cabana F, Page C, Svotelis A, Langlois-Michaud S, Tousignant M. Is an in-home telerehabilitation program for people with proximal humerus fracture as effective as a conventional face-to face rehabilitation program? A study protocol for a noninferiority randomized clinical trial. BMC Sports Sci Med Rehabil. 2016 Aug 26;8(1):27. doi: 10.1186/s13102-016-0051-z. eCollection 2016. PMID 27570627